CLINICAL TRIAL: NCT06509477
Title: A Randomized, Double-masked, Active Controlled, Within-subject Equivalency Clinical Trial to Compare Effectiveness and Safety of Lunaphil Ultra (Hyaluronic Acid, Produced by Espad Pharmed Co.) Versus Juvederm Ultra 4® (Hyaluronic Acid, Produced by Allergan Co.) for the Management of Moderate or Severe Nasolabial Folds
Brief Title: Effectiveness and Safety Comparison of Lunaphil Ultra (Hyaluronic Acid, by Espad Pharmed Co.) Versus Juvederm Ultra 4® (Hyaluronic Acid, by Allergan Co.) in Nasolabial Folds (NLFs) Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUN.ESP.KB.IV.00
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Moderate or Severe Nasolabial Folds
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-masked, active controlled, within-subject, paired, and equivalency clinical trial. Subjects were treated with Lunaphil Ultra in one NLF and Juvederm Ultra 4® in the opposite NLF.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lunaphil Ultra (by Espad Pharmed Co.) (Experimental): Lunaphil Ultra (by Espad Pharmed Co.) will be administered over a 2-week period (initial treatment plus one touch-up) to achieve optimal correction of the NLFs. In case of suboptimal correction of NLFs at week 2 after the initial treatment, the treating investigator will be directed to retreat the under corrected NLF(s).
  Interventions: Device: Hyaluronic acid Lunaphil Ultra (by Espad Pharmed Co.)
- Juvederm Ultra 4® (by Allergan Co.) (Active Comparator): Juvederm Ultra 4® (by Allergan Co.) will be administered over a 2-week period (initial treatment plus one touch-up) to achieve optimal correction of the NLFs. In case of suboptimal correction of NLFs at week 2 after the initial treatment, the treating investigator will be directed to retreat the under corrected NLF(s).
  Interventions: Device: Hyaluronic acid Juvederm Ultra 4® (by Allergan Co.)

INTERVENTIONS:
Device: Hyaluronic acid Lunaphil Ultra (by Espad Pharmed Co.) — Two treatments will be allowed over a 2-week period (initial treatment plus one touch-up) to achieve optimal correction of the NLFs based on investigator's opinion
  Arms: Lunaphil Ultra (by Espad Pharmed Co.)
Device: Hyaluronic acid Juvederm Ultra 4® (by Allergan Co.) — Two treatments will be allowed over a 2-week period (initial treatment plus one touch-up) to achieve optimal correction of the NLFs based on investigator's opinion
  Arms: Juvederm Ultra 4® (by Allergan Co.)

SUMMARY:
Rationale and background: Skin aging is a complex process that results in various changes in the skin, including wrinkles, sun spots, and sagging skin. The NLF is a natural change that becomes more prominent with aging and significantly affects the beauty of the facial skin. Dermal fillers, particularly hyaluronic acid (HA) fillers, are commonly used to correct these signs of aging. This study aimed to compare the effectiveness and safety of Lunaphil Ultra with Juvederm Ultra 4® for treating NLFs.

Primary objective: Effectiveness assessment of Lunaphil Ultra Secondary objectives: Effectiveness and safety assessment of Lunaphil Ultra Study design: This is a randomized, double-masked, active controlled, within-subject, and equivalency clinical trial.

Setting: Subjects were treated with Lunaphil Ultra in one NLF and Juvederm Ultra 4® in the opposite NLF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 30 years of age
* Visible bilateral NLFs that were approximately symmetrical and had an equal severity ranging from moderate to severe (assessed at the deepest part)
* Able to follow study instructions and likely to complete all required visits
* Signed informed consent

Exclusion Criteria:

* History of bleeding disorders or participants receiving or recently exposed (≤ 3 weeks) to continuous treatment with thrombolytics, anticoagulants, platelet inhibitors, or NSAIDs
* Acute herpetic eruption
* Known susceptibility to keloid formation, hypertrophic scarring or clinically significant skin pigmentation disorders
* Known sensitivity to local anesthetics of the amide type (such as lidocaine), history of hypersensitivity to gram-positive bacterial proteins, history of multiple severe allergies, history of anaphylactic shock
* Known hypersensitivity to any component of the study products or excipients (like hyaluronic acid)
* History of receiving immune therapy or a history of autoimmune disease
* History of active chronic debilitating systemic disease
* History of connective tissue disease, history of malignancy (except for non-melanoma skin cancer) within the last 5 years
* Clinically significant active dermatologic disorders within the last 6 months
* Use of oral retinoids, over-the-counter (OTC) or prescription antiwrinkle treatments, microdermabrasion, or chemical peels in the NLF area within the last 4 weeks or intention to use them during the study
* Any prior cosmetic procedure or tissue augmentation at the NLF injection site within 1 year before study entry (or intent to undergo such a procedure during the study)
* Pregnancy or breastfeeding

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Balighi, Prof. Derm, Principal Investigator — Department of Dermatology, Razi Hospital, Tehran University of Medical Sciences, Tehran, Iran.
Locations (1):
- Orchid Pharmed, Medical Department, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: NLF
Groups:
- Group 1: Each participant received Lunaphil Ultra on right NLF and Juvederm Ultra 4® on the left NLF
- Group 2: Each participant received Lunaphil Ultra on left NLF and Juvederm Ultra 4® on the right NLF
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 52; 104 NLF | 52; 104 NLF
Lunaphil Ultra | 52; 52 NLF | 52; 52 NLF
Juvederm Ultra 4® | 52; 52 NLF | 52; 52 NLF
Completed | 51; 102 NLF | 46; 92 NLF
Not Completed | 1; 2 NLF | 6; 12 NLF

BASELINE CHARACTERISTICS:
Groups:
- Total Participants: Each participant received Lunaphil Ultra on one NLF and Juvederm Ultra 4® on the other NLF
Arm/Group | Total Participants
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.39 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Level of Improvement From Baseline in NLF Severity Score by Wrinkle Severity Rating Scale (WSRS)
Description: The scores are from 1 to 5, 1 indicating no visible folds and 5 indicating extreme folds
Time Frame: 24 weeks
Population: 29 participants were excluded from the per-protocol (PP) population due to protocol violation; In addition, 4 participants with missing data at week 24 and 4 participants with missing data at week 12 (for imputation) were excluded from the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
Number analyzed (Participants) | 100 | 100
score on a scale
  PP population: number analyzed (Participants) | 75 | 75
  PP population | -0.80 (0.66) | -0.81 (0.67)
  ITT population | -0.73 (0.66) | -0.74 (0.67)
Statistical Analysis 1: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); ITT population; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.01 to 0.03], Standard Deviation 0.10
Statistical Analysis 2: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); PP population; Test type: Other; p > 0.99, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.013 to 0.040], Standard Deviation 0.11

2. Secondary Outcome: Number of Subjects With an Improved Score From Baseline Based on Physician Global Aesthetic Improvement Scale (PGAIS)
Description: The scores are from 1 to 5, 1 indicating exceptional improvement and 5 indicating worsened results
Time Frame: 24 weeks
Population: ITT Population; 7 participants with missing data at week 24 were excluded from the intention-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
Number analyzed (Participants) | 97 | 97
Participants
  Assessor 1 | 66 | 66
  Assessor 2 | 79 | 79
Statistical Analysis 1: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); Assessor1; Test type: Other; p > 0.99, McNemar
Statistical Analysis 2: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); Assessor 2; Test type: Other; p > 0.99, McNemar

3. Secondary Outcome: Number of NLFs Maintaining a Clinically Significant Improvement in NLF Severity Score by Wrinkle Severity Rating Scale (WSRS)
Description: ≥1-point reduction from baseline. The scores are from 1 to 5, 1 indicating no visible folds and 5 indicating extreme folds
Time Frame: 24 weeks
Population: ITT population; 74 NLF in each group had clinically significant improvement in NLF severity score by Wrinkle Severity Rating Scale (WSRS)
Measure: Count of Units; unit: NLF
Units Other Than Participants: NLF
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
Number analyzed (Participants) | 74 | 74
Number analyzed (NLF) | 74 | 74
NLF | 43 | 43
Statistical Analysis 1: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); Test type: Other; p > 0.99, McNemar

4. Secondary Outcome: The Injected Volume to Obtain Optimal Aesthetic Result
Description: initial treatment + touch-up
Time Frame: 2 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
Number analyzed (Participants) | 104 | 104
cc | 0.90 (0.29) | 0.88 (0.29)
Statistical Analysis 1: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); Test type: Other; p = 0.49, t-test, 2 sided

5. Secondary Outcome: The Number of NLFs Receiving Touch-up Treatment
Description: Counting the number of NLF who need additional injection
Time Frame: 2 weeks
Population: ITT population
Measure: Count of Units; unit: NLF
Units Other Than Participants: NLF
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
Number analyzed (Participants) | 104 | 104
Number analyzed (NLF) | 104 | 104
NLF | 74 | 69
Statistical Analysis 1: Comparison: Lunaphil Ultra (by Espad Pharmed Co.) vs Juvederm Ultra 4® (by Allergan Co.); Test type: Other; p = 0.33, McNemar

6. Secondary Outcome: Evaluation of Adverse Events During 24 Weeks
Description: All reported AEs are classified based on the Medical Dictionary for Regulatory Activities (MedDRA) terms and are graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: 24 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
Number analyzed (Participants) | 104 | 104
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Lunaphil Ultra (by Espad Pharmed Co.) | Juvederm Ultra 4® (by Allergan Co.)
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 3/104 | 5/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lunaphil Ultra (by Espad Pharmed Co.) (N=104) | Juvederm Ultra 4® (by Allergan Co.) (N=104)
Injection site erythema (General disorders) | 2 | 0
Injection site pain (General disorders) | 1 | 1
Injection site swelling (General disorders) | 1 | 2
Injection site mass (General disorders) | 0 | 1
Injection site nodule (General disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT06509477/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT06509477/SAP_001.pdf